CLINICAL TRIAL: NCT03725111
Title: Haemodynamics Variations of Transcutaneous Oxygen in Patient With Arterio-venous Leg Ulcers Under Venous Compression (COMPULCE Study)
Brief Title: Haemodynamics Variations of Transcutaneous Oxygen in Patient With Areterio-venous Leg Ulcers Under Venous Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A01048-47
Record Dates: First submitted 2018-10-19; First posted 2018-10-30 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2018-11

CONDITIONS: Leg Ulcer; Compression; Vein
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- arterio venous leg ulcers (Experimental)
  Interventions: Device: venous compression

INTERVENTIONS:
Device: venous compression — venous compression

SUMMARY:
Arterio-venous leg ulcers are real problems when it comes to public health because it has a major cost and leads to social and professional handicap.

The management of leg ulcers is not clear and can be venous compression or surgery.

The aim of the study is to evaluate the variation of the transcutaneous oxygen with compression.

The second aim is to see how tolerate is the compression and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* age eighteen or more
* leg arteio-venous ulcers

Exclusion Criteria:

* age Under eighteen,
* Index pressure in the ankle Under 0.5

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
haemodynamic variation of the transcutaneous oxygen | 1 month
  measurement of the transcutaneous oxygen during two different appointement using a transcutaneous monitor TCM4

CONTACTS AND LOCATIONS:
Locations (1):
- ELHOMSY, Caen, Basse Normandie, France